CLINICAL TRIAL: NCT04315012
Title: The Effect of E-mobile Education on The Quality of Life in Breast Cancer Women
Brief Title: Training With Mobile Application in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Derya ÇINAR, Asistant Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bakircay University
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; quality of life; endocrine hormonal therapy; mobile phone; mobil app; education of patients; smartphone
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The data were collected to with face to face and/or telephone interviews at 2 time points: prior to the initiation (T0) and after the completion (T1) of mobile app-based education. Mobile application was including information about breast cancer definition, treatment process, symptoms management, adequate nutrition, regular physical activity and coping with stress. In this process, the control group patients were provided with standard care
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving mobile app-based education (Experimental): to receive mobile app-based education on quality of life of women diagnosed with breast cancer implementation of adjuvant endocrine hormonal therapy.
  Interventions: Other: receive mobile app-based education
- Standart (No Intervention): not to receive mobile app-based education on quality of life of women diagnosed with breast cancer implementation of adjuvant endocrine hormonal therapy.

INTERVENTIONS:
Other: receive mobile app-based education — to receive mobile app-based education on quality of life of women diagnosed with breast cancer implementation of adjuvant endocrine hormonal therapy.
  Arms: Receiving mobile app-based education

SUMMARY:
Endocrine hormonal therapy (EHT) applied to avoid recurrence and metastasis of the breast cancer has also side effects which do not threaten life; however, it does negatively effects quality of life. The objective of this study was to determine the effects on quality of life of a mobile app-based (e-mobile) education for supportive care of patients with breast cancer receiving adjuvant endocrine hormonal therapy. The data were collected to with face to face and/or telephone interviews at 2 time points: prior to the initiation (T0) and after the completion (T1) of mobile app-based education. Patients were received education via mobile app for 12 weeks during which they were contacted in every 15 days; a mobile app-based (e-mobile) education was provided, including information about breast cancer definition, treatment process, symptoms management, adequate nutrition, regular physical activity and coping with stress. In this process, the control group patients were provided with standard care.

DETAILED DESCRIPTION:
Mobile devices have an increasing role for the patient care and its use in the field of oncology creates promising opportunities for supportive cancer care and patient education. Mobile applications were established for the supportive cancer care but their area of use is limited. Although there are many field specific medical mobile applications, there are few training programs for the benefit of patients. However, these are innovative tools and provide accessibility, individual training and consultancy in order for the patients to be able to cope with side effects of the treatment; thus, improving their quality of life, symptom management and distress.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary breast cancer,
* Non-metastatic,
* Hormone receptor positive (ER positive and/or PR positive)
* For whom adjuvant EHT was implemented at least for three months

Exclusion Criteria:

* Diagnosed with secondary breast cancer,
* Metastatic,
* Hormone receptor negative (ER negative and/or PR negative)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Functional Assessment for the Cancer Treatment - Endocrine Symptoms Quality of Life Scale (FACT-ES QLS) | Change from Baseline Quality of Life at 12 weeks
  The scale includes five sub dimensions and total of 46 items measuring the well-being of patients within the course of the last 7 days. There are sub dimensions for each of the following: physical well-being (7 items, 0-28 points), social/family well-being (7 items, 0-28 points), emotional well-being (6 items, 0-24 points), functional well-being (7 items, 0-28 points) and endocrine symptoms (19 items, 0-76 points). Endocrine symptoms' subdimension contains symptoms related to the side effects of EHT. The range of total points of the scale is 0-184. It shows that quality of life increases as total points of the scale increase. It shows that quality of life decreases as total points of the scale decrease.
National Comprehensive Cancer Network (NCCN) Distress Thermometer | Change from Baseline Distress at 12 weeks
  Patients may specify the severity of the distress level they experienced related to their problems, with these numbers, within the course of last 7 days. No distress is specified with "0" point, a severe amount of distress is specified with "10" points.

CONTACTS AND LOCATIONS:
Overall Officials: DERYA ÇINAR, Principal Investigator — İzmir Bakırçay University
Locations (1):
- İzmir Bakırçay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No